CLINICAL TRIAL: NCT03982134
Title: Phase Ib Study to Assess Safety and Tolerability of PDR001 in Combination With Panobinostat in Metastatic Melanoma and Non-small Cell Lung Cancer After Failure of Prior Anti PD1 or PD-L1 Therapy
Brief Title: PDR001 + Panobinostat for Melanoma and NSCLC
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision to withdraw
Sponsor: Muhammad Furqan (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Muhammad Furqan, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201904832
Record Dates: First submitted 2019-06-06; First posted 2019-06-11 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Melanoma; Non Small Cell Lung Cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung | interventions — spartalizumab; Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PDR001 with Panobinostat (Experimental): All enrolled patients will be treated with a combination of PDR001 at 400mg every 4 weeks and panobinostat. Dose and frequency of Panobinostat will vary depending upon the dose-level cohort of the study participants. Each participant will be assigned to a particular dose-level cohort.
  Interventions: Drug: PDR001; Drug: Panobinostat

INTERVENTIONS:
Drug: PDR001 — PDR001 is a humanized IgG4 antibody
  Other Names: spartalizumab
Drug: Panobinostat — Panobinostat is a Histone deacetylase inhibitor (HDACi).
  Other Names: LBH589 lactate

SUMMARY:
The purpose of this research study is to find the dose of the study drug PDR001 that, when given in combination with the drug Panobinostat, results in the best outcomes for metastatic melanoma and non-small cell lung cancer (NSCLC)

DETAILED DESCRIPTION:
This is an open label, non-randomized Phase Ib study combining PDR001 with HDAC inhibitor Panobinostat in patients with metastatic melanoma and NSCLC who have failed prior Anti PD1 or PD-L1 therapy.

The primary purpose of this study is to find the recommended Phase II dose (RP2D) of Panobinostat in combination with PDR001. Standard 3+3 design will be used for dose escalation or de-escalation. Depending upon tolerability and dosing, the total number of participants may vary from 9-24. Initially patients will start from dose level '0' and there will be 1 dose escalation level '1' and two de-escalation levels ('-1' and '-2'). The maximum number in each dose level will be 6.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study have to meet all of the following criteria:

* Patients must provide written informed consent prior to any screening procedures.
* Age 18 years or older.
* Willing and able to comply with scheduled visits, treatment plan and laboratory tests
* Able to swallow and retain oral medication Panobinostat
* Histologically or cytologically confirmed diagnosis of melanoma or NSCLC
* ECOG performance status of 0-2
* Patients with melanoma and NSCLC must have progressed clinically as determined by the treating physician on a prior line of anti-PD-1/PD-L1 therapy. If they have received more than one line of prior therapy, the last treatment must be with an anti-PD-1/PDL-1 inhibitor, alone or in combination with another systemic therapy (e.g. chemotherapy, CTLA4 inhibitor).
* Patients with NSCLC who are known to have targetable genomic alterations (including EGFR exon 19 deletion or L858R substitution, ALK rearrangement, ROS1 fusion, NTRK 13 fusions, BRAF V600 mutation), must have progressed on or could not tolerate FDA approved targeted therapy for the alterations mentioned above, in addition to progressed on PD-1/L1 Checkpoint blockade to be eligible for the study. Patients with Melanoma who are known to have BRAF V600 mutation must have progressed on or could not tolerate BRAF-targeted therapy with or without MEK inhibitor in addition to PD-1/PD-L1 checkpoint inhibitor to be eligible for the study.

Exclusion Criteria:

Patients eligible for this study must not meet any of the following criteria:

* Presence of symptomatic central nervous system (CNS) metastases, or CNS metastases that require local CNS-directed therapy (such as radiotherapy or surgery), or increasing doses of corticosteroids within the prior 2 weeks. Patients with residual symptoms that are either controlled or improving after treatment will be allowed to participate in the study.
* History of severe hypersensitivity reactions to other mAbs
* Prior treatment with an HDAC inhibitor
* Patients who meet the following laboratory criteria:

Hematology:

* Neutrophil count of </=1500/mm3
* Platelet count of </=100,000/mm3
* Hemoglobin < 8 g/dL (Transfusion support is allowed to meet the eligibility)

Biochemistry:

* AST/SGOT and ALT/SGPT >3 x upper limit of normal (ULN) or > 5.0 x ULN if the transaminase elevation is due to disease involvement
* Serum bilirubin > 1.5 x ULN
* Creatinine clearance (calculated using Cockcroft-Gault formula, or measured) </=40 mL/min
* Impaired cardiac function or clinically significant cardiac disease, including any of the following:

  * Clinically significant and/or uncontrolled heart disease such as congestive heart failure requiring treatment (NYHA grade >/= 2), uncontrolled hypertension or clinically significant arrhythmia
  * Corrected QT (QTcF) > 450 msec for males and females using Fridericia's correction on screening ECG or congenital long QT syndrome
  * Acute myocardial infarction or unstable angina pectoris < 3 months prior to study entry
  * Presence of any clinically significant cardiac arrhythmias, e.g. ventricular, supraventricular, nodal arrhythmias, or conduction abnormality
  * Left Ventricular Ejection Fraction (LVEF) < 40%, as determined by echocardiogram (ECHO) or Multiple Gated acquisition (MUGA)
  * Subjects with active, known or suspected autoimmune disease requiring systemic immunosuppression. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
  * History of drug-induced pneumonitis
  * Active infection requiring systemic antibiotic therapy.
  * Known history of Human Immunodeficiency Virus (HIV) infection.
  * Known history of active HBV or HCV infection. Testing for HBV or HCV status is not necessary unless clinically indicated or the patient has a history of HBV or HCV infection.
  * Unresolved diarrhea ≥ CTCAE grade 2 or presence of medical condition associated with chronic diarrhea (such as irritable bowel syndrome, inflammatory bowel disease).
  * Malignant disease, other than that being treated in this study. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within 2 years prior to study treatment; completely resected basal cell and squamous cell skin cancers; any malignancy considered to be indolent and that has never required systemic chemo or immunotherapy therapy (e.g. ductal carcinoma in situ, some low grade lymphomas, high-grade prostatic intraepithelial neoplasia, monoclonal gammopathy of undetermined significance); and completely resected carcinoma in situ of any type.
  * Any condition that would prevent the patient's participation in the clinical study due to safety concerns, compliance with clinical study procedures or interpretation of study results.
  * Systemic anti-cancer therapy within 2 weeks of the first dose of study treatment. For cytotoxic agents that have major delayed toxicity, e.g. mitomycin C and nitrosoureas, 4 weeks is indicated as washout period. For patients receiving anticancer immunotherapies such as CTLA-4 antagonists, 3 weeks is indicated as the washout period
  * Patients requiring chronic treatment with systemic steroid therapy, other than replacement dose steroids in the setting of adrenal insufficiency. Topical, inhaled, nasal and ophthalmic steroids are allowed.
  * Patients receiving systemic treatment with any immunosuppressive medication (other than steroids as described above). Patients with prior history of allogeneic organ transplant will be excluded.
  * Use of any live vaccines within 4 weeks of initiation of study treatment.
  * Major surgery within 2 weeks of the first dose of study treatment (mediastinoscopy, insertion of a central venous access device, and insertion of a feeding tube are not considered major surgery).
  * Patient who has received thoracic radiotherapy to lung fields ≤ 4 weeks prior to starting the study treatment or patients who have not recovered from radiotherapy-related toxicities to CTCAE grade ≤1 (except alopecia and lymphopenia). For all other anatomic sites (including radiotherapy to thoracic vertebrae and ribs) radiotherapy ≤ 2 weeks prior to starting the study treatment or has not recovered from radiotherapy-related toxicities to CTCAE grade ≤1 (except alopecia and lymphopenia). Palliative radiotherapy for bone lesions ≤ 2 weeks prior to starting study treatment is allowed.
  * Participation in an interventional, investigational study within 2 weeks of the first dose of study treatment.
  * Presence of ≥ CTCAE grade 2 toxicity (except alopecia, regardless of grade), lymphopenia, peripheral neuropathy and ototoxicity, which are excluded if ≥ CTCAE grade 3) due to prior anti-cancer therapy.
  * Use of hematopoietic colony-stimulating growth factors (e.g. G-CSF, GMCSF, M-CSF) ≤2 weeks prior start of study drug. An erythroid stimulating agent is allowed as long as it was initiated at least 2 weeks prior to the first dose of study treatment.
  * Pregnant or lactating women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 150 days after the last dose of PDR001. Highly effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male sterilization (at least 6 months prior to screening). For female patients on the study the vasectomized male partner should be the sole partner for that patient.
  * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
  * In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
  * Women are considered post-menopausal and not of child bearing potential if they have had over 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile age appropriate (e.g. generally 40-59 years), history of vasomotor symptoms (e.g. hot flushes) in the absence of other medical justification or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
* Sexually active males unless they use a condom during intercourse while taking the study treatment and for 150 days after stopping study treatment and should not father a child in this period. A condom is required to be used also by vasectomized men as well as during intercourse with a male partner in order to prevent delivery of the drug via seminal fluid.
* Concomitant use of strong CYP3A4 inducers (Carbamazepine, Modafinil, Rifampin, Rifabutin, Rifapentin, Phenytoin, Phenobarbital and St. John's wort) or strong inhibitors like Cimetidine, Grapefruit juice and Seville oranges as mentioned in appendix E. If patient can come off of these drugs and receive an alternative therapy then they will be eligible as far as time equals 4 half-lives of that medication has elapsed prior to starting protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of PDR001 in combination with panobinostat in determining a recommended Phase II dose | Initiation of treatment up to 2 years
  The recommended Phase 2 dose will be determined by using a 3 + 3 design with 1 dose escalation and 2 dose deescalation cohorts. Safety assessments will consist of monitoring and recording all adverse events, including serious adverse events, the monitoring of hematology, chemistry, ECG and the regular monitoring of vital signs, thyroid function, pregnancy and physical exam including weight and performance status.

SECONDARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) using CTCAE, Version 5.0 | Initiation of treatment up to 2 years
  All adverse events (AEs) will be considered in DLT assessment unless the event is clearly unrelated to trial treatment. The National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 will be used.
Progression free survival (PFS) per RECIST 1.1 | Initiation of treatment up to 2 years
  PFS is defined as the time between the first dose of study therapy and the earliest date of progression or death (participants who have neither progressed nor dies will be censored at the most recent last-known-alive date).
Overall survival (OS) | Initiation of treatment up to 2 years
  OS is calculated from time when study therapy begins to death from any cause.
Overall Response Rate (ORR) per RECIST 1.1 | Initiation of treatment up to 2 years
  OS is defined as the time between the first dose of study therapy and death (participants who have not died will be censored at the most recent last-known-alive date).

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Furqan, MD, Principal Investigator — University of Iowa

IPD SHARING:
Plan to Share IPD: No